CLINICAL TRIAL: NCT06219330
Title: "Salivary Levels of Cathelicidin LL-37 in Patients With Oral Potentially Malignant Lesions, A Case Control Study"
Brief Title: Cathelicidin LL-37 Relation to Potentially Malignant Lesions
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Sandy Hassan, Associate professor oral medicine & periodontology departement, Fayoum University
Other Study IDs: 63723
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Oral Potentially Malignant Lesions
Keywords: Oral potentially malignant lesions, Cathelicidin LL-37

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (control group): 15 Healthy participants without any oral lesions
- Group II:: 15 Patients having atrophic/erosive oral lichen planus (OLP). Group III: 15 Patients having oral leukoplakia
- Group III:: 15 Patients having oral leukoplakia

SUMMARY:
LL-37 appears to have a potential role in potentially malignant lesions (OLP & leukoplakia). The remarkable diagnostic accuracy of salivary LL-37 in differentiating potentially malignant lesion and healthy control could confirm its utilization as an innovative marker to early diagnose potentially malignant lesions. Salivary LL-37 being non-invasive accurate marker could be as a chair-side diagnostic method that detect potentially malignant lesions.

DETAILED DESCRIPTION:
Aim: The recognition of practical early diagnostic biomarkers is a cornerstone of improved prevention and treatment of cancer thus the current study estimated salivary level of Cathelicidin LL-37 in patients suffering from potentially malignant lesions and control subjects to corroborate Cathelicidin LL-37 as a diagnostic marker for early detection of potentially malignant diseases and revealing its possible role in carcinogenesis.

Methodology: 45 systemically healthy individuals were subdivided into three groups: Group I: 15 Healthy participants without any oral lesions. Group II: 15 Patients having atrophic/erosive oral lichen planus (OLP). Group III: 15 Patients having oral leukoplakia.. Enzyme linked immune-sorbent assay (ELIZA) kit was used to evaluate the level of LL-37 in whole unstimulated salivary samples collected from all participants. To reveal AUC, sensitivity, specificity, and diagnostic accuracy of LL-37 receiver operating curve (ROC) analysis was done.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age range 30 - 70 years.
* Patients agreed to sign a written consent after understanding the nature of the study.
* Clinically diagnosed and histologically confirmed as having oral potentially malignant lesions mainly atrophic/erosive oral lichen planus and oral leukoplakia.

Exclusion Criteria:

* Systemic diseases as well as pregnant or lactating females.
* Patients currently taking corticosteroids, immunosuppressives drugs, contraceptive pills, or antibiotics.
* Patients are diagnosed with any other oral lesions other than oral lichen planus and oral leukoplakia.
* Vulnerable subjects as prisoners, or mentally disabled.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of 45 systemically healthy participants were included in this study that were divided equally into 3 groups: Group I: 15 Healthy participants without any oral lesions. Group II: 15 Patients having atrophic/ erosive oral lichen planus. Group III: 15 Patients having oral leukoplakia.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Cathelicidin LL-37 level in salivary samples from all participants mesured using ELISA | level of LL-37 is measured after the completion of all sample collection carried at the 1 day of enrollement of subjects in the investigation after diagnosis confirmation
  ELISA is used to estimate Cathelicidin LL-37 levels in saliva samples from patients with OPMD compared to healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Sandy hassan shaaban, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No